CLINICAL TRIAL: NCT02841137
Title: Effect of Progesterone 5, 10, and 20 mg Tablets Compared To Progesterone 100 mg Capsules on the Endometrial Thickness of Post-Menopausal Women Under Hormone Therapy - A Prospective, Open-Label, Randomized, Four-Arm, Parallel-Group, Phase II Clinical Trial
Brief Title: Efficacy Study of Progesterone Tablet in Post-menopausal Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: IBSA Institut Biochimique SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16CDN-Prg02
Record Dates: First submitted 2016-07-14; First posted 2016-07-22 (Estimated); Last update posted 2018-06-11 (Actual); Status verified 2017-08

CONDITIONS: Menopause
MeSH Terms: interventions — Progesterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- progesterone 5 mg (Experimental): progesterone 5 mg tablet
  Interventions: Drug: Progesterone
- progesterone 10 mg (Experimental): progesterone 10 mg tablet
  Interventions: Drug: Progesterone
- progesterone 20 mg (Experimental): progesterone 20 mg tablet
  Interventions: Drug: Progesterone
- progesterone 100 mg (Active Comparator): progesterone 100 mg capsule
  Interventions: Drug: Progesterone

INTERVENTIONS:
Drug: Progesterone — comparison of different dosages of drug towards the active comparator

SUMMARY:
This is a phase II study intended to determine the effect of progesterone 5, 10 and 20 mg tablets compared to progesterone 100 mg capsules on the endometrial thickness of post-menopausal women under hormone therapy with estradiol.

ELIGIBILITY:
Inclusion Criteria:

1. Availability for the entire study period
2. Post-menopausal female defined as:

   * at least 12 consecutive months of spontaneous amenorrhea and
   * less than 10 years of spontaneous amenorrhea, and
   * Follicle-stimulating hormone (FSH) levels > 40 milli International Units/ml
3. Females with an intact uterus
4. Moderate to severe climacteric vasomotor symptoms
5. Aged of at least 40 years but not older than 65 years
6. Body mass index (BMI) greater than or equal to 18.00 kg/m2 and below 30.00 kg/m2
7. Non- or ex-smoker;
8. Endometrium thickness ≤4 mm on ultrasonography at screening
9. Negative mammogram (dated < 2 years)
10. Negative Pap smear test (dated < 1 year)
11. Normal clinical breast examination
12. Normal pelvic examination
13. Have no clinically significant diseases captured in the medical history or evidence of clinically significant findings on physical examination, as determined by the medical investigator
14. Willingness to adhere to the protocol requirements as evidenced by the informed consent form (ICF) duly read, signed and dated by the subject

Exclusion Criteria:

1. Use of any estrogen, progestin, or estrogen/progestin drug products, androgens, selective estrogen receptor modulators (SERMs), phytoestrogen supplements or natural products (soy, black cohosh, dong quai) during the past 3 months before the screening visit
2. Use of any estrogen, progestin or androgen pellet or injectable therapy during the past 6 months before the screening visit
3. Contraindications to hormone therapy:

   * Active liver dysfunction or disease or history of severe liver disease
   * Known, suspected or past history of hepatic tumors (benign or malign)
   * Active or past history of arterial thromboembolic disease (e.g. angina, myocardial infarction, stroke, coronary heart disease, transient ischemic attack)
   * Active or past history of venous thromboembolism (e.g. deep venous thrombosis, pulmonary embolism) or active thrombophlebitis
   * Known, suspected or past history of breast cancer
   * Known, suspected or past history of estrogen-dependent or progestin-dependent malignant neoplasia (e.g. endometrial cancer)
   * Endometrial hyperplasia
   * Porphyria cutanea tarda
   * Genital bleeding
   * Untreated hypertension
   * Classical migraine
   * Partial or complete loss of vision or diplopia due to ophthalmic vascular disease
4. Presence of clinically significant screening ECG abnormalities as defined by medical judgment
5. Presence of polyps
6. Presence of uterine fibroids or other abnormalities affecting endometrial thickness measurement or precluding estrogen therapy
7. Known hypersensitivity to the active substances or to any of the excipients contained in the drug products in particular to soya or peanut, as well as hereditary problems of fructose intolerance or phenylketonuria
8. Participation in a concurrent clinical trial or another trial within the past 2 months
9. Use of any enzyme-modifying drugs, including strong inhibitors of cytochrome P450 (CYP) enzymes (such as cimetidine, fluoxetine, quinidine, erythromycin, ciprofloxacin, fluconazole, ketoconazole, diltiazem and HIV antivirals) and strong inducers of CYP enzymes (such as barbiturates, carbamazepine, glucocorticoids, phenytoin, rifampin and St John's Wort), in the previous 28 days before day 1 of this study
10. Maintenance therapy with any drug or significant history of drug dependency, drug abuse or alcohol abuse within the last 2 years
11. Presence of any medical condition or other circumstances which would significantly decrease the chance of obtaining reliable data, achieving study objectives or completing the study
12. Serious psychiatric problems (whether or not receiving treatment) or in any case such as to compromise the patient's reliability
13. Any clinically significant illness in the previous 28 days before day 1 of this study
14. Any history of tuberculosis and/or prophylaxis for tuberculosis
15. Positive screening of alcohol and/or drugs of abuse
16. Positive results to HIV Ag/Ab combo, hepatitis B surface antigen or hepatitis C virus tests
17. Females who are pregnant according to a positive serum pregnancy test
18. Presumption of subject's poor reliability/cooperation
19. Any reason which, in the opinion of the Investigator, would prevent the subject from participating in the study

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-06; Primary Completion 2017-08-02 (Actual); Study Completion 2018-04-25 (Actual)

PRIMARY OUTCOMES:
endometrial thickness change towards baseline (mm) | 3 months

SECONDARY OUTCOMES:
histological assessment of the endometrium (presence of hyperplasia or proliferation) | 3 months
bleeding (presence or absence) | everyday over 3 months
quality of life (MENQOL Questionnaire) | 3 months
sleep scale from the Medical Outcomes Study (MOS) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Deschamps, Principal Investigator — Algorithme Pharma Inc
Locations (1):
- Algorithme Pharma, Mount Royal, Quebec, Canada